CLINICAL TRIAL: NCT06457659
Title: Effect of Early Prosthetic Fitting in Patients With Below Knee Amputation
Brief Title: Effect of Early Prosthetic Fitting in Patients With Below-knee Amputation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/728
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Amputation Stump

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Rehab Group (Experimental)
  Interventions: Behavioral: Early Rehab Group
- Delayed Rehab Group (Other)
  Interventions: Other: Delayed Rehab Group

INTERVENTIONS:
Behavioral: Early Rehab Group — The first group of 25 Patients was fitted with Prosthesis with in 6months of duration after amputation. The basic theme was to check the physical psychological and QOL in early prostheic-fitted patients through WHO_QOL.
  Arms: Early Rehab Group
Other: Delayed Rehab Group — The 2nd group of 25 patients was fitted with Prosthesis after 6 months after amputation. No physical rehab was done during this period including physiotherapy and prosthetic treatment. The main aim was to check the significant impact of delayed rehabilitation.
  Arms: Delayed Rehab Group

SUMMARY:
A randomized control trial of 50 patients to identify the effect of early prosthetic fitting and physical rehabilitation. Previous studies show a significant impact of early induction of prosthetic rehabilitation of amputation. Delayed rehabilitation may cause severe physical complications like joint contracture, and muscle strength loss.

DETAILED DESCRIPTION:
Along with physical complications delays in rehabilitation may also significantly affect psychological, economic, and quality of daily life. Pakistan is a low-income developed country and the major cause of amputation here is traumatic amputation, which affects mostly younger age people. After missing a precious body part if the amputee comes along with such kind of physical and Psychological complications, his/her whole daily life will be affected. There is a keen need for the implementation of global rules for physical rehabilitation of amputees and disabled including the duration of induction of prosthetics as well as overall physical rehabilitation after surgical and traumatic removal of limbs.

ELIGIBILITY:
Inclusion Criteria:

* Male and female below-knee amputees due to trauma and diabetes were included

Exclusion Criteria:

* patients with comorbidities and old users of prostheses were excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
World Health Organization Quality of life (WHO QOL) | 12 Months
  Questionnaire was used to measure the impact in both groups on quality of life. The WHOQOL is a quality-of-life assessment developed by the WHOQOL Group with fifteen international field centers, simultaneously, in an attempt to develop a quality-of-life assessment that would be applicable cross-culturally. The patient's physical, psychological, social, and environmental state of health is assessed separately in WHO_QOL known as the 4 domains of the questionnaire. 0 points represent the worst possible state of health, while 100 points represent the best possible state of health about the respective domain.

CONTACTS AND LOCATIONS:
Locations (1):
- Mobility Rehab care, Islamabad Medical Center, Dera Ismail Khan, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No